CLINICAL TRIAL: NCT02270619
Title: Sleep Loss as a Vulnerability Factor for Inflammation Induced Depressive Symptoms in Older Women
Brief Title: Sleep Health, Inflammation, and Emotion Study
Acronym: SHINE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Hyong Jin Cho, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: K23AG049085 (NIH)
Record Dates: First submitted 2014-10-15; First posted 2014-10-21 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Endotoxins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Uninterrupted sleep & placebo (Placebo Comparator): Uninterrupted sleep followed by placebo
  Interventions: Other: Placebo; Other: Uninterrupted sleep
- Uninterrupted sleep & endotoxin (Experimental): Uninterrupted sleep followed by endotoxin 0.8 ng/kg of body weight IV bolus
  Interventions: Biological: Endotoxin; Other: Uninterrupted sleep
- Partial sleep deprivation & placebo (Experimental): Partial sleep deprivation followed by placebo
  Interventions: Behavioral: Partial sleep deprivation; Other: Placebo
- Partial sleep deprivation & endotoxin (Experimental): Partial sleep deprivation followed by endotoxin 0.8 ng/kg of body weight IV bolus
  Interventions: Biological: Endotoxin; Behavioral: Partial sleep deprivation

INTERVENTIONS:
Biological: Endotoxin — Low dose endotoxin (0.8 ng/kg of body weight) as IV bolus
  Arms: Partial sleep deprivation & endotoxin; Uninterrupted sleep & endotoxin
Behavioral: Partial sleep deprivation — Partial night sleep deprivation by staying awake from 23:00 to 03:00
  Arms: Partial sleep deprivation & endotoxin; Partial sleep deprivation & placebo
Other: Placebo — 0.9% saline as IV bolus
  Arms: Partial sleep deprivation & placebo; Uninterrupted sleep & placebo
Other: Uninterrupted sleep — Uninterrupted sleep from 23:00 to 07:00
  Arms: Uninterrupted sleep & endotoxin; Uninterrupted sleep & placebo

SUMMARY:
Late-life depression is a major public health burden due to its high prevalence and associated morbidity, suicide risk, functional decline, and mortality. Unfortunately, current antidepressant therapies have limited effectiveness; hence, biologically plausible models for new treatments are being pursued. Systemic inflammation is hypothesized to play an important role on the onset and perpetuation of depression, especially in older women. Aging processes involve a heightened inflammatory state, and both inflammatory disorders and depression are more prevalent in women than men. However, increased systemic inflammation does not necessarily lead to depression in all women. Even when robust systemic inflammation is experimentally induced (e.g. endotoxin administration), largely variable increases in depressive symptoms are found. Defining the factors that account for this variability may identify individuals at risk of developing depression when exposed to heightened inflammatory states such as aging, obesity, and chronic disease, and informs future translational studies of depression prevention. In particular, the role of sleep disturbance in explaining this variability requires further attention because it is an independent risk factor for depression and heightens systemic inflammation by increasing the production of proinflammatory cytokines. The investigators have also discovered that women, but not men, who report sleep disturbance including short sleep duration experience significantly more depressive symptoms in response to an inflammatory challenge than women without sleep disturbance. Thus, it is hypothesized that sleep loss is a vulnerability factor for inflammation-induced depressive symptoms in women. However, to date, no experimental approach has been used to evaluate the role of sleep loss on inflammation-induced depressive symptoms. This proposal aims to examine this hypothesis by partial sleep deprivation (PSD) followed by endotoxin challenge in older women. It also aims to explore genomic and socio- emotional mechanisms underlying the association between sleep loss and depressive symptoms. In a randomized controlled factorial design, 80 healthy female volunteers aged 60 to 80 will be randomly assigned to one of 4 arms: 1) uninterrupted sleep followed by placebo; 2) uninterrupted sleep followed by endotoxin; 3) PSD followed by placebo; or 4) PSD followed by endotoxin. Subjects will be administered placebo or endotoxin in the morning after PSD or uninterrupted sleep. Depressive symptoms will be repeatedly assessed over 6 hours after placebo or endotoxin administration.

ELIGIBILITY:
Inclusion Criteria:

* to be in good general health
* to be female
* to be aged 60 to 80 years

Exclusion Criteria:

* presence of chronic mental or physical illnesses
* history of allergies, auto-immune, liver, or other chronic diseases
* current use of prescription medications such as steroids, non-steroid anti-inflammatory drugs, immune modifying drugs, opioid analgesics, and psychotropic medications
* current sleep disorders such as insomnia or sleep apnea
* nightshift work or time zone shifts (> 3 hours) within the previous 6 weeks
* an Axis I psychiatric disorder as determined by the Research Version of the Structured Clinical Interview for DSM-5 (SCID-5-RV) including a current or within 1 year prior-to-study history of major depressive disorder (a history of depression 1 or more years prior to the study is not an exclusion criterion, which will be considered for a pre-planned sensitivity analysis, however, any prior depressive episode severe enough to have involved suicidal ideation or required an inpatient psychiatric admission is an exclusion criterion)
* prior or current suicidal ideation assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
* current depressive symptoms assessed by the Patient Health Questionnaire (PHQ-9) (≥ 5)
* sleep disorders identified by the SCID and the Duke Structured Interview for Sleep Disorders (DSISD)
* sleep disturbance defined by the Pittsburgh Sleep Quality Index (PSQI) (≥ 5)
* a positive screen for sleep apnea using the Berlin Sleep Apnea Questionnaire
* excessive caffeine use (>600 mg/day)
* BMI > 35 due to the effects of obesity on cytokine activity and risk for sleep disordered breathing
* evidence of recreational drug use from urine test
* any abnormalities on screening laboratory tests.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-10; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms from baseline | At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after drug administration
  Short Form of the Profile of Mood States (POMS-SF)

SECONDARY OUTCOMES:
Change in fatigue from baseline | At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after drug administration
  Short Form of the Profile of Mood States (POMS-SF)
Change in pain from baseline | At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after drug administration
  Modified Pennebaker Inventory of Limbic Languidness (PILL) and Visual Analogue Scale (VAS)
Anhedonia | 2 hours after drug administration
  Facial expressions and skin conductance in response to funny film clips

OTHER OUTCOMES:
Change in proinflammatory cytokines from baseline | At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after drug administration
  Circulating proinflammatory cytokines ((interleukin-1 receptor antagonist, interleukin-6, tumor necrosis factor-α, and soluble tumor necrosis factor receptor)
Change in gene expression from baseline | At baseline and then at 30 minutes after drug administration
  Genome-wide transcriptional profiling; Expression of genes involved in proinflammatory pathways and in circadian clock network

CONTACTS AND LOCATIONS:
Overall Officials: Hyong Jin Cho, MD, PhD, Principal Investigator — University of California, Los Angeles; Michael R Irwin, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Cousins Center for Psychoneuroimmunology, Los Angeles, California, United States